CLINICAL TRIAL: NCT04499482
Title: Safety and Tolerability of Soy Fiber in the Elderly: A Dose Escalation Study
Brief Title: Safety and Tolerability of Soy Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Candida Rebello, Assistant Professor, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PBRC 2020-010; 1K99AG065419-01A1 (NIH)
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Safety Issues; Tolerance
MeSH Terms: interventions — Food

STUDY DESIGN:
Intervention Model Description: Dose escalating cross over trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foods containing 10 g soy flour (Experimental): Participants will receive foods containing 10 g of soy flour to be consumed everyday for one week. If they tolerate the dose, they will receive the next dose without any wash-out period.
  Interventions: Other: Food
- Foods containing 20 g soy flour (Experimental): Participants will receive foods containing 20 g of soy flour to be consumed everyday for one week. If they tolerate the dose, they will receive the next dose without any wash-out period.
  Interventions: Other: Food
- Foods containing 30 g soy flour (Experimental): Participants will receive foods containing 30 g of soy flour to be consumed everyday for one week.
  Interventions: Other: Food

INTERVENTIONS:
Other: Food — Soy-fiber containing food

SUMMARY:
This is a dose escalation trial in the elderly with obesity to determine the maximum tolerated dose of a novel dietary fiber from whole young soy pods (soy) delivered in foods.

DETAILED DESCRIPTION:
The tolerability to 10 g, 20 g, and 30 g of soy will be tested. At each dose, eight subjects will incorporate the foods containing soy into their usual diet for one week. The tolerability to each dose will be evaluated and fecal short chain fatty acids will be measured as a biomarker of compliance. Subjects who satisfy the eligibility criteria and express willingness to consume the study foods will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Adult (70 - 85 years).
* Body mass index between 30 and 40 kg/m2.
* No evidence of diabetes (fasting blood sugar <126 mg/dL).
* No evidence of dementia (MMSE score > 25).
* No evidence of depression. (Geriatric Depression Scale-15 [GDS-15] < 6.
* Are weight stable (< 3 kg weight change in the past three months).

Exclusion Criteria:

* Have type 1 or type 2 diabetes currently being treated by medication.
* Report clinically significant gastrointestinal malabsorption syndromes such as chronic diarrhea, or celiac disease.
* Are being treated with medications that have a significant effect on insulin resistance, obesity, and metabolic rate, or medications that significantly increase body weight such as antidepressants, second-generation antipsychotics, systemic glucocorticoids, and adrenergic blockers or stimulators (unless the dose and body weight have been stable for six months).
* Have serum triglyceride concentrations > 400 mg/dl.
* Clinically significant abnormal laboratory markers (as determined by the medical investigator).
* Subjects with anticipated surgery during the study period.
* Subjects with a reported history of substance abuse or alcoholism or significant psychiatric disorder that would interfere with the ability to complete the study.
* Subjects who are current smokers or have smoked within the previous three months. Smoking is not permitted during the study.
* Subjects who are unable to provide a baseline blood or fecal sample or if they have any condition that impedes testing of the study hypothesis or makes it unsafe to consume the food being tested in the study (determined by the investigative team).
* Women on hormone replacement therapy unless weight has been stable over the last six months.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candida Rebello, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 8 subjects. Each subject started at the 10g soy flour dose and crossed over to the 20 g soy flour dose after one week if they tolerated the 10 g soy flour dose, and subsequently to the 30g soy flour dose if they tolerated the 20g soy flour dose.
Groups:
- Foods Containing 10 g Soy Flour: Participants will receive foods containing 10 g of soy flour to be consumed everyday for one week.
  Food: Soy-fiber containing food
Period: Foods Containing 10 g Soy Flour
Arm/Group | Foods Containing 10 g Soy Flour
Started | 8
Completed | 7
Not Completed | 1
Not completed — One subject dropped from the study at Day 3 as the subject could not meet the demands of the study | 1
Period: Foods Containing 20 g Soy Flour
Arm/Group | Foods Containing 10 g Soy Flour
Started | 7
Completed | 7
Not Completed | 0
Period: Foods Containing 30g Soy Flour
Arm/Group | Foods Containing 10 g Soy Flour
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The participant dropped from the study was excluded from the analysis. The data relates to seven participants who were tested for tolerance to the three doses of soy flour
Groups:
- All Study Participants: Participants will receive foods containing 10g, 20g, and 30g of soy flour to be consumed everyday for one week at each dose.
  Food: Soy-fiber containing food
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: One subject dropped from the study at day 3 of week one and was not included in the analysis
  Years | 73 (2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject dropped from the study at Day 3 of week one and was not included in the analysis
  Participants
    Female | 3
    Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject dropped from the study at Day 3 of week one and was not included in the analysis.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 2
    White | 5
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: Each of the seven subjects crossed over to the next treatment
  participants
    United States | 7
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Each of the seven subjects crossed over to the next treatment
  kg/m^2 | 34 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events Following Each Dose of Soy
Description: Dose safety will be investigated by compiling by treatment (e.g. 10 g dose, 20 g dose, 30 g dose) a list of adverse events such as frequency of headaches, nausea, vomiting. The study physician in consultation with the coordinator will review and determine safety
Time Frame: One week at each dose
Population: One subject dropped from the study at Day 3 of week one and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Foods Containing 20 g Soy Flour: Participants will receive foods containing 20 g of soy flour to be consumed everyday for one week.
  Food: Soy-fiber containing food
Arm/Group | Foods Containing 10 g Soy Flour | Foods Containing 20 g Soy Flour | Foods Containing 30 g Soy Flour
Number analyzed (Participants) | 7 | 7 | 7
Participants | 0 | 1 | 1

2. Primary Outcome: 10 g Soy-related Gastrointestinal Symptoms
Description: Subjects will complete a gastrointestinal symptoms questionnaire. The ratings are none, mild, moderate, and severe.
Time Frame: One week
Population: One subject dropped from the study at Day 3 of week one and was excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 10 g Soy Flour
Number analyzed (Participants) | 7
Participants
  Bloating: Mild | 1
  Bloating: None | 6
  Abdominal Rumbling: Mild | 2
  Abdominal Rumbling: None | 5
  Flatulence: Mild | 2
  Flatulence: None | 5
  Abdominal Pain: Mild | 0
  Abdominal Pain: None | 7

3. Primary Outcome: 20 g Soy-related Gastrointestinal Symptoms
Description: Subjects will complete a gastrointestinal symptoms questionnaire. The ratings are none, mild, moderate, and severe.
Time Frame: One week
Population: One subject dropped out of the study on Day 3 of Week 1 and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 20 g Soy Flour
Number analyzed (Participants) | 7
Participants
  Bloating: Mild | 0
  Bloating: None | 7
  Abdominal Rumbling: Mild | 1
  Abdominal Rumbling: None | 6
  Flatulence: Mild | 5
  Flatulence: None | 2
  Abdominal pain: Mild | 0
  Abdominal pain: None | 7

4. Primary Outcome: 30 g Soy-related Gastrointestinal Symptoms
Description: Subjects will complete a gastrointestinal symptoms questionnaire. The ratings are none, mild, moderate, and severe.
Time Frame: One week
Population: One subject dropped out of the study on Day 3 of Week 1 and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 30 g Soy Flour
Number analyzed (Participants) | 7
Participants
  Bloating: Mild | 1
  Bloating: None | 6
  Abdominal Rumbling: Mild | 1
  Abdominal Rumbling: None | 6
  Flatulence: Mild | 5
  Flatulence: None | 2
  Abdominal Pain: Mild | 1
  Abdominal Pain: None | 6

5. Primary Outcome: 10 g Soy-related Stool Frequency
Description: Subjects will complete the stool frequency questionnaire. Stool frequency will be rated from 0 to more than 9 over three consecutive days in each week
Time Frame: One week
Population: One subject dropped out of the study on Day 3 of Week 1 and was not included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 10 g Soy Flour
Number analyzed (Participants) | 7
Participants
  1-2 | 2
  3-4 | 4
  5-6 | 1

6. Primary Outcome: 20 g Soy-related Stool Frequency
Description: as for outcome 5
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 20 g Soy Flour
Number analyzed (Participants) | 7
Participants
  1-2 | 1
  3-4 | 5
  5-6 | 1

7. Primary Outcome: 30 g Soy-related Stool Frequency
Description: as for outcome 5
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 30 g Soy Flour
Number analyzed (Participants) | 7
Participants
  1-2 | 1
  3-4 | 3
  5-6 | 3

8. Primary Outcome: 10 Soy-related Stool Consistency
Description: Subjects will complete a stool consistency questionnaire. Stool consistency will be rated according to the Bristol Stool Scale where scores from three to five will be considered normal and 1, 2, 6, and 7 will be considered abnormal.
Time Frame: One week
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 10 g Soy Flour
Number analyzed (Participants) | 7
Participants
  3, Normal (Like sausage but with cracks) | 2
  4, Normal (Like sausage, smooth and soft | 3
  5, Normal (Soft blobs with clear cut edges) | 2
  1, Abnormal(Separate hard lumps) | 0
  2, Abnormal (Sausage-shaped but lumpy) | 0
  6, Abnormal (Fluffy pieces with ragged edges) | 0
  7, Abnormal (Watery) | 0

9. Primary Outcome: 20 g Soy-related Stool Consistency
Description: as for outcome 8
Time Frame: One week
Population: One subject was dropped from the study on Day 3 of week 1 and was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 20 g Soy Flour
Number analyzed (Participants) | 7
Participants
  3, Normal (Like a sausage, but with cracks) | 0
  4, Normal (Like sausage, smooth and soft) | 5
  5, Normal (Soft blobs with clear-cut edges) | 2
  1, Abnormal (Separate hard lumps) | 0
  2, Abnormal (Sausage-shaped but lumpy) | 0
  6, Abnormal (Fluffy pieces with ragged edges) | 0
  7, Abnormal (Watery) | 0

10. Primary Outcome: 30 g Soy-related Stool Consistency
Description: as for outcome 8
Time Frame: One week
Population: One subject was dropped from the study at Day 3 and was not included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Foods Containing 30 g Soy Flour
Number analyzed (Participants) | 7
Participants
  3, Normal (Like a sausage but with cracks) | 0
  4, Normal (Like a sausage, smooth and soft) | 2
  5, Normal (Soft blobs with clear-cut edges) | 4
  1, Abnormal (Separate hard lumps) | 1
  2, Abnormal (Sausage-shaped but lumpy) | 0
  6, Abnormal (Fluffy pieces with ragged edges) | 0
  7, Abnormal (Watery) | 0

11. Secondary Outcome: 10 g Soy Intake Effect on Fecal Short Chain Fatty Acids
Description: Measurement of fecal short chain fatty acids in response to intake of soy
Time Frame: One week
Population: One subject was dropped from the study at Day 3 and was excluded from the analysis
Measure: Mean (Standard Error); unit: mg fecal short chain fatty acids/g dry f
Arm/Group | Foods Containing 10 g Soy Flour
Number analyzed (Participants) | 7
mg fecal short chain fatty acids/g dry f | 5736.93 (1615.02)

12. Secondary Outcome: 20 g Soy Intake Effect on Fecal Short Chain Fatty Acids
Description: Measurement of fecal short chain fatty acids in response to intake of soy
Time Frame: One week
Population: One subject was dropped from the study at Day 3 and was excluded from the analysis.
Measure: Mean (Standard Error); unit: mg fecal short chain fatty acids/g dry f
Arm/Group | Foods Containing 20 g Soy Flour
Number analyzed (Participants) | 7
mg fecal short chain fatty acids/g dry f | 6577.87 (1615.02)

13. Secondary Outcome: 30 g Soy Intake Effect on Fecal Short Chain Fatty Acids
Description: Measurement of fecal short chain fatty acids in response to intake of soy
Time Frame: One week
Population: One subject was dropped from the study at Day 3 and was excluded from the analysis
Measure: Mean (Standard Error); unit: mg fecal short chain fatty acids/g dry f
Arm/Group | Foods Containing 30 g Soy Flour
Number analyzed (Participants) | 7
mg fecal short chain fatty acids/g dry f | 6191.89 (1615.02)

ADVERSE EVENTS:
Time Frame: One week at each dose
Groups:
- Foods Containing 10g Soy Flour: Participants will receive foods containing 10 g of soy flour to be consumed everyday for one week.
  Food: Soy-fiber containing food
- Foods Containing 20g Soy Flour: Participants will receive foods containing 20 g of soy flour to be consumed everyday for one week.
  Food: Soy-fiber containing food
- Foods Containing 30g Soy Flour: Participants will receive foods containing 30 g of soy flour to be consumed everyday for one week.
  Food: Soy-fiber containing food
Arm/Group | Foods Containing 10g Soy Flour | Foods Containing 20g Soy Flour | Foods Containing 30g Soy Flour
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 1/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Foods Containing 10g Soy Flour (N=8) | Foods Containing 20g Soy Flour (N=7) | Foods Containing 30g Soy Flour (N=7)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Mild flatulence
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — Mild constipation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT04499482/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT04499482/ICF_001.pdf